CLINICAL TRIAL: NCT01942941
Title: Prospective Observational Series to Establish the Haemodynamic Efficacy and Tolerability of gekoTM Device in Patients With Lower Limb Vascular Disease
Brief Title: Peripheral Vascular Disease and Nerve Stimulation
Acronym: CCLINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/EE/0314
Record Dates: First submitted 2013-09-04; First posted 2013-09-16 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Critical Limb Ischaemia; Claudication; Ulcers; Varicose Veins; Post Angioplasty
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Intermittent Claudication; Ulcer; Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- geko™ electrical stimulation (Experimental): Applied to stimulate peroneal nerve unilaterally
  Interventions: Device: geko™ electrical stimulation

INTERVENTIONS:
Device: geko™ electrical stimulation — applied to stimulate peroneal nerve and cause active muscle twitch

SUMMARY:
A study to see what effect the geko™ device has on blood flow in patients with lower limb vascular disease.

DETAILED DESCRIPTION:
The geko™ device, (CE 558928; British Standards Institute notified body 0086),is a wearable, discrete, self-contained stimulation unit that adheres to the skin (see www.gekodevices.com). The, geko™ triggers small electrical impulses that gently activate the common peroneal nerve within the popliteal fossa, behind the knee, in turn activating the venous muscle pumps of the calf and foot. Substantive increases in lower limb blood flow have been demonstrated to improve arterial, venous and microcirculatory blood flow with no reported morbidity.

Environmental Conditions The examinations will be carried out in a designated temperature controlled clinical room in the Vascular Lab at Hull Royal Infirmary. Participants will be required to abstain from vigorous exercise, nicotine, caffeine and fatty foods prior to their examination. They will be required to wear light garments with their legs exposed.

The geko™ device will be applied to outer/ posterior aspect of the knee whilst the subjects are semi-recumbent, with their knees flexed. The participants will be given 30 minutes in the quiet, environmentally controlled room prior to commencement of measurement to enable equilibration.

Assessments Participants will complete the McGill Pain questionnaire prior to device activation Participants will have the geko™ device applied whilst semi-recumbent with their knees flexed. The intensity will be increased until visible muscle stimulation is evident (concentric isotonic contractions) or until patient tolerance is reached

* Laser Doppler imaging will be used to assess microcirculation flow on the dorsum of both feet at:

  1. Baseline (rest)
  2. 5 minute intervals while the geko™ device is active
  3. 30 minutes following removal of the device Laser Doppler flowmetry is a reproducible, objective, non-invasive measurement which can be used to evaluate real time cutaneous blood flow. The low powered light is conducted via glass fibres to a probe attached to the skin and is scattered by the movement of blood cells inducing a Doppler shift. This allows information on flux and cell velocity to be recorded. The system to be used for this trial is the Moor Instruments DT-4 mains unit with integrated bilateral lasers.
* Ultrasound Doppler arterial flow velocity and blood volume flow within the femoral artery (mid thigh) bilaterally at:

  1. Baseline (rest)
  2. 30 minutes while the device is active
* Ultrasound Doppler flow velocity in femoral vein (mid thigh) bilaterally at:

  1. Baseline (rest)
  2. 40 minutes while the geko is active
* Vascular Endothelial Growth Factor (VEGF), Tissue Plasminogen Activator antigen (TPA antigen), Full blood count (FBC) and Plasminogen activator inhibitor-1 (PAI-1): 15 mls of blood to be taken from both femoral veins at:

  1. Baseline (rest)
  2. 45 minutes while the geko™ device is active ELISA analysis will be carried out on samples (see appendix). Vascular Endothelial Growth Factor - Therapies which can lead to the development of new, collateral blood vessels, are of particular interest in the field of peripheral arterial disease where narrowing or blockages in existing blood vessels result in tissue ischaemia. Vascular endothelial growth factor (VEGF) is a signal protein produced by cells that stimulates the growth of new blood vessels from pre-existing vessels. Several previous studies have shown that electrical stimulation increases VEGF levels and in turn increases vessel density in muscles.

Tissue plasminogen activator (tPA) is a protein involved in the breakdown of blood clots. As a result it has therapeutic uses in clinical medicine to treat thromboses and emboli. Electrical stimulation has been previously shown to provoke an acute release of tPA into the circulation, although it appears that this response decreases with repeated stimulations. Use of the geko™ device has been shown to result in a significant decrease in Tissue Plasminogen Activator (tPA) antigen which is indicative of increased fibrinolytic activity.

Plasminogen activator inhibitor- 1 (PAI-1) is the primary inhibitor of plasminogen activators and inactivates tissue plasminogen activator (t-PA) and urokinase-type plasminogen activator (u-PA). PAI-1 is an important inhibitor of the fibrinolytic system, and elevated levels could suppress fibrinolysis and result in an increased risk of thrombosis. Increased PAI-1 levels have been shown to be associated with a number of atherosclerotic risk factors, PAI-1 has been shown to act as a prothrombic factor in both arterial and venous thromboembolic disorders.

* Ankle Brachial Pressure Index at baseline and post removal of geko™- utilising both Posterior Tibial Artery and Anterior Tibial Artery
* Maximum calf circumference at baseline and post removal of geko™
* Three blood pressure and heart rate measurements will be taken bilaterally at baseline and @ 30 minutes while the device is active. The mean of the three values will be used for comparison.
* Patient tolerance/ acceptability + Nurse tolerance/ ease of application Questionnaire using Visual Analogue Scores and Verbal Rating Scores to be completed following removal of geko™ device (see appendix)
* The McGill Pain Questionnaire to be completed following device removal

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Absence of haematological disorders or DVT (deep vein thrombosis) in the preceding 12 months
* Intact cutaneous sensations to nocioception in the lower limb, as determined by the investigator
* Intact healthy skin at site of application
* On effective contraception if sexually active - oral contraceptive pill (> 3 months use), condoms, intrauterine contraceptive device, depot injection
* Able to understand the Patient Information Sheet and capable and willing to give informed consent and follow the protocol requirements

Exclusion Criteria:

* History of haematological disorder or DVT in the preceding 12 months
* Pregnant or planning to become pregnant during study duration
* Pacemakers or implantable defibrillators
* Use of any other neuro-modulation device
* Current use of TENS (transcutaneous electrical nerve stimulation) in pelvic region, back or legs
* Use of investigational drug/device therapy within past 4 weeks that may interfere with this study.
* Significant varicose veins or lower limb ulceration.
* Recent surgery (such as abdominal, gynaecological, hip knee replacement).
* Recent trauma to lower limbs.
* Chronic Obesity (BMI Index >34).
* Any medication judged to be significant by the Principal Investigator.
* Any significant illness during the four (4) weeks preceding the screening period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Effect of geko™ on blood volume flow through the femoral artery | Study day i.e. 1 day
  Measured with ultrasound doppler

SECONDARY OUTCOMES:
Effect of geko™ on venous blow flow | Study day i.e. 1 day
  Measured with ultrasound doppler
Effect of geko™ on microcirculatory flow | Study day i.e. 1 day
  Measured with laser doppler
Establish whether effects of geko™ are local or systemic | Study day i.e. 1 day
  Measurements will be taken from both the leg on which the device is active and the leg with no geko™
Effect of geko™ on patients symptoms | study day i.e. 1 day
  Completion of McGill pain questionnaire and visual analogue scale
Acceptability and tolerability of geko™ device | study day i.e. 1 day
  Completion of tolerability questionnaire
Effect of gekoTM on calf circumference | Study day i.e. 1 day
  Calf circumference measured before and after device

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Barnes, MRCS, MA, Principal Investigator — Academic Department of Vascular Surgery, Hull Royal Infirmary/ Hull York Medical School
Locations (1):
- Hull Royal Infirmary, Hull, EastRiding of Yorkshire, United Kingdom